CLINICAL TRIAL: NCT02140437
Title: An Open-label, Multi-center, Randomized Phase II Study of Fulvestrant Anastrozole Combination Versus Anastrozole Alone in Patients With Luminal A-like Postmenopausal Advanced Breast Cancer
Brief Title: Fulvestrant Combined Anastrozole Versus Anastrozole in Luminal A-like Postmenopausal ABC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The progress of enrollment is too slow.
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xichun Hu, M.D. Ph. D., Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fudan BR2014-14
Record Dates: First submitted 2014-05-09; First posted 2014-05-16 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Carcinoma Breast Stage IV
Keywords: Fulvestrant; Anastrozole; Luminal A-like; Postmenopausal; Advanced breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant; Anastrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fulvestrant and anastrozole (Experimental): Anastrozole 1 mg PO QD Fulvestrant 500mg IM d1,15, 29 and 4 weeks after
  Interventions: Drug: Fulvestrant; Drug: Anastrozole
- Anastrozole (Active Comparator): Anastrozole 1 mg PO QD
  Interventions: Drug: Anastrozole

INTERVENTIONS:
Drug: Fulvestrant — Adding fulvestrant to the standard endocrine therapy, anastrozole
  Other Names: falsodex
  Arms: Fulvestrant and anastrozole
Drug: Anastrozole — standard endocrine therapy
  Other Names: Arimidex

SUMMARY:
This research is designed to investigate whether the addition of fulvestrant 500mg to anastrozole is better than anastrozole alone as first-line endocrine therapy for advanced breast cancer.

DETAILED DESCRIPTION:
Anastrozole is the standard first-line endocrine treatment for patients with hormonal receptor positive advanced breast cancer. It has been proven that the addition of fulvestrant 250mg can enhance PFS of anastrozole monotherapy according to SWOG0226 study. However, the optimal recommended dose of fulvestrant for patients with advanced breast cancer is 500mg worldwide according to CONFIRM study. The investigator designed this research to investigate whether high dose fulvestrant can further improve efficacy of anastrozole monotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Histologically confirmed breast cancer
3. Luminal A-like breast cancer (primary or metastatic tumor), defined as: ER-positive, PR-positive (> 20%), Her-2 negative and Ki67 <14%.
4. Advanced breast cancer is eligible:

   * Endocrine therapy-naive patients with locally advanced disease, who are not suitable for radical surgery or radiotherapy (the decision made by the multidisciplinary breast cancer team). Prior first-line cytotoxic chemotherapy is acceptable. or
   * Patients with recurrent or metastatic disease, who have not received adjuvant endocrine therapy or who have been 2 years or longer after stop of adjuvant endocrine therapy. Patients who had disease progression from first-line cytotoxic chemotherapy are allowed.
5. At least one lesion (measurable and / or non-measurable) can be assessed at baseline, and is suitable for repeated assessments with CT and/or MRI.
6. Postmenopausal women, defined as any one of the following criteria (as defined in the NCCN's menopause definition):

   * previous bilateral oophorectomy
   * 60 years old or older
   * less than 60 years old, amenorrheic for 12 months or longer in the absence of chemotherapy, tamoxifen, toremifene, or ovarian suppression and follicle-stimulating hormone and estradiol in the postmenopausal range.
   * If taking tamoxifen, or toremifene and age < 60, then FSH and E in the postmenopausal range
7. ECOG 0, 1 or 2.
8. Patients with good compliance.
9. Must be able to swallow tablets.
10. Without any significant gastrointestinal obstruction or dysfunction of absorption for oral drug.

Exclusion Criteria:

1. Life-threatening metastatic visceral disease, defined as extensive liver involvement or any degree of brain or leptomeningeal involvement (past or present) or symptomatic pulmonary lymphatic metastasis. If the investigator believe that their respiratory function is not significantly impaired due to illness, patients with scattered parenchymal metastases are qualified.
2. Have received any systemic treatment other than first-line cytotoxic chemotherapy.
3. Radiation therapy within 28 days prior to randomization (exception: radiotherapy to control bone pain, but should be completed before the randomization).
4. Use any other anti-cancer therapy at the same time (except bisphosphonate).
5. Previous endocrine treatment for advanced breast cancer.
6. Current or previous malignancy ( except for breast cancer, basal cell or squamous cell carcinoma of the skin with adequate treatment, cervical carcinoma in situ).
7. Inadequate blood or liver or renal function within one week prior to randomization: Platelets < 80 × 10^9/L; Total bilirubin > 1.5 × (ULRR) (patients with Gilbert's syndrome is eligible); or ALT or AST > 2.5 × ULRR (without liver metastases) or > 5 × ULRR (with liver metastases).
8. History with hemorrhagic constitution (e.g. disseminated intravascular coagulation, clotting factor deficiency) or long-term anticoagulant therapy.
9. Hypersensitivity history to excipients or castor oil of fulvestrant or anastrozole.
10. Any other severe co-existing medical disorders, ie uncontrolled heart disease.
11. Participation in any clinical trial and / or exposure to any investigational medication within 28 days before randomization.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2015-12 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
PFS(Progression free survival) | 8 weeks

SECONDARY OUTCOMES:
OS(overall survival ) | 8 weeks

OTHER OUTCOMES:
ORR(objective response rate) | 8 weeks
CBR(Clinical benefit rate) | 8 weeks
Number of patients with grade 3 or 4 adverse events | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xichun Hu, MD.PhD., Principal Investigator — Fudan University